CLINICAL TRIAL: NCT06217991
Title: A Single-center, Prospective, Single-arm Clinical Study of Laparoscopic Proximal Gastrectomy Based on an Original Esophagogastric Anastomose (PTST,Parachute- Tunnel- Style Technique)
Brief Title: A Clinical Study of Laparoscopic Proximal Gastrectomy Based on PTST(Parachute-tunnel- Style Technique) Esophagogastric Anastomose.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XKT-Y-20221148
Record Dates: First submitted 2023-12-17; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Gastroesophageal-junction Cancer; Proximal Gastrectomy; Gastroesophagostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PTST anastomose group after proximal gastrectomy (Experimental): Standard procedure: Patient placed in a supine position and proximal gastrectomy performed under general anesthesia.
  1. Lymph node dissection
  2. Cut the esophagus
  3. Gymnosis of gastric curvature greater and gastric curvature lesser
  4. The specimen removed from the stomach(5cm away)
  5. Preparation of serosa-muscle flap: Mark two straight lines, A and B, about 3cm long, with methylene blue on the anterior wall of the stomach about 2cm and 6cm from the gastric stump. The electrocoagulation and cutting power of the electrotome were adjusted to 10 watts, and the serosa-muscle layer of the gastric wall was cut along the marked line with the electrotome. With the help of the assistant, the surgeon separated the gastric parietal serosa-muscle layer from the submucosa along line B to line A. When the dissociation reached the middle point of the tunnel, it should be dissociated along line A to line B, completely dissociated the gastric parietal serosa-muscle layer from the submucosa.
  Interventions: Procedure: PTST(parachute-tunnel-style technique)for esophagogastrostomy

INTERVENTIONS:
Procedure: PTST(parachute-tunnel-style technique)for esophagogastrostomy — Suture the gastric remnant at the mark on the back wall of the esophagus.(Don't tighten the suture); Pull the esophageal stump out of the tunnel meanwhile tighten the suture and the gastric stump to close the back wall of the esophagus and the gastric stump together;Cut the back esophageal wall close to the esophageal stump,cut the front gastric wall along line B. Suture the back esophageal wall and the upper edge of the front gastric wall incision from right to left;Remove residual esophageal nail, and suture the back esophageal wall and the lower edge of the gastric incision from right to left. Suture the anterior wall of the stomach at the lower edge of the tunnel with the serosa layer at the lower edge of the front wall of the esophagus stomach anastomosis;Suture the upper edge of the tunnel with the front wall of the esophagus and the left and right lateral walls at the gastric stump suture of the original posterior wall of the esophagus. (all use 3-0 barbed suture continuously)

SUMMARY:
1. To evaluate the safety, simplicity and effectiveness of the gastric function (anti-reflux) preservation of the innovative "parachute-tunnel-style technique" (PTST) in laparoscopic proximal gastrectomy.
2. To investigate the correlation between anastomotic stenosis and blood supply of serosa-muscle flap,suture after esophagogastric anastomosis.(obtain objective indexes such as blood supply, healing pattern and length change of serosa-muscle flap through animal experiments)

ELIGIBILITY:
Inclusion Criteria:

* Gastric cancer was confirmed histopathologically;
* Patients who may undergo proximal gastrectomy according to guidelines;
* Early upper gastric cancer, more than 1/2 of the distal gastric remnant remained after resection;
* Esophagogastric junction carcinoma with maximum diameter ≤4 cm;
* Patients with advanced upper gastric cancer (MSI-H) achieved cCR by neoadjuvant immunochemotherapy.

Exclusion Criteria:

* Patients with systemic conditions that cannot tolerate laparoscopic surgery;
* Distal gastric remnant was less than 1/2 after proximal gastrectomy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
occurrence rate of anastomotic stenosis | one month after surgery
  morbidity(%)
occurrence rate of reflux esophagitis | three month after surgery; six month after surgery
  * Visick score after surgery
  * Los Angeles rating

CONTACTS AND LOCATIONS:
Locations (1):
- General Surgery Gastrointestinal Department,Tang-Du of Fourth Military Medical University, Xi'an, Shannxi Province, China